CLINICAL TRIAL: NCT06480760
Title: Effects of Carnosine In Patients With Peripheral Arterial Disease Patients; Randomized Intervention Trial (CIPHER)
Brief Title: Effects of Carnosine In Patients With Peripheral Arterial Disease Patients
Acronym: CIPHER
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Shahid Baba (Other)
Collaborators: National Institutes of Health (NIH) (NIH); National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Sponsor-Investigator, Shahid Baba, Professor, University of Louisville
Organization: University of Louisville (Other)
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 24.0309; R01HL163419 (NIH)
Record Dates: First submitted 2024-06-24; First posted 2024-06-28 (Actual); Last update posted 2025-05-29 (Actual); Status verified 2025-05

CONDITIONS: Peripheral Arterial Disease
Keywords: peripheral arterial disease; carnosine
MeSH Terms: conditions — Peripheral Arterial Disease | interventions — Carnosine

STUDY DESIGN:
Intervention Model Description: A randomized, double-blinded longitudinal study in approximately 144 PAD patients
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Placebo (No Intervention): Cellulose
- Carnosine (Experimental): Carnosine 2 g daily for 6 months
  Interventions: Drug: Carnosine

INTERVENTIONS:
Drug: Carnosine — Food ingredient (supplement)
  Arms: Carnosine

SUMMARY:
The purpose of this study is to determine whether carnosine (a food ingredient found in chicken and red meat) supplementation (2 g) for 6 months in participants with non-claudication and claudication peripheral arterial disease (PAD) improves walking ability. Previous studies with heart failure patients have shown that carnosine supplementation increases walking capacity in these patients.

DETAILED DESCRIPTION:
The objective of this double-blinded longitudinal study is to determine whether carnosine supplementation (2 g) for 6 months in participants with non-claudication and claudication peripheral arterial disease (PAD) improves walking ability. In this pilot study we will enroll 144 participants that will be divided into placebo (n=72) and carnosine groups (n=72). We will measure the distance covered on the 6-minute walk test (6-MWT) and the pain free walking capacity on the treadmill before and after the placebo or carnosine supplementation. We will measure ankle branchial index (ABI) and blood flow by magnetic resonance imaging (MRI) before and after the carnosine and placebo supplementation. In addition, we will measure carnosine by 1HMRS (Proton magnetic resonance spectroscopy), perform, global metabolomics and proteomics in the skeletal muscle, a comprehensive lipid and metabolic profile of blood, uptake of carnosine in red blood cells (RBCs), and measure carnosine aldehyde conjugates in the urine before and after 6 months of carnosine and placebo supplementation. Following completion of the study, we will follow the participants for another 3 months and examine the durability of carnosine supplementation.

ELIGIBILITY:
Inclusion Criteria:

1. Participants between 40-80 years of age.
2. White or African American race.
3. Literate in English.
4. ABI >0.4-<0.90, obtained within 6 weeks from enrollment.
5. Willing and able to comply with protocol requirements.
6. Participant is able to provide informed consent.

Exclusion Criteria:

1. As per physician's discretion, participants with HIV, hepatitis, significant liver disease, anemia, renal disease requiring dialysis, lung disease requiring home oxygen therapy, and active cancer may be excluded.
2. Critical limb ischemia with below or above the knee amputations or any form of foot ulceration over the symptomatic leg.
3. Presence of significant injury within 30 days, or vascular intervention on the symptomatic leg within 6 months before enrollment, as per physician's discretion.
4. Participants with a baseline 6MWT of less than 152.0 meters (498ft) or greater than 487.7 meters (1600ft).
5. Known allergy to L-carnosine.
6. Participants with rare autosomal recessive metabolic disorder carnosinemia or carnosinase deficiency.
7. Currently participating in other clinical trials.
8. Participation in any carnosine supplementation clinical trial anytime in the past.
9. Participants already taking carnosine.
10. Participants unable to provide urine sample (anuric).
11. Pregnant participants.
12. Participants using dual antiplatelet therapies will not be included for biopsy.
13. Participants with internal metallic objects in body will not be eligible for MRI or 1HMRS.

Ages: 40 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 144 (Estimated)
Dates: Start 2025-05-20 (Actual); Primary Completion 2028-10-01 (Estimated); Study Completion 2028-10-01 (Estimated)

PRIMARY OUTCOMES:
Measure distance covered on six-minute walk test (6MWT) | Baseline, 3 months, 6 months, 9 months
  Distance covered on a flat and hard surface in 6 minutes. Units: Feet

SECONDARY OUTCOMES:
Measure Ankle-Brachial Index (ABI) | Baseline, 3 months, 6 months, 9 months
  Ratio of blood pressure measurements from the arms and ankles. Units: Normal range 1.0-1.4 and lower than 0.9 is an indication of peripheral arterial disease
Treadmill Testing | Baseline, 3 months, 6 months
  Graded treadmill testing using the Gardener protocol until the onset of the maximal claudication pain.
  Units: Meters
Skin Integrity | Baseline, 3 months, 6 months
  Check the color, trophic changes and flakes. Units: None
Musculoskeletal Assessment | Baseline, 3 months, 6 months
  Perform goniometric measurements, assess pain and conduct muscle strength testing. Upper limb muscle strength will be evaluated by hand-grip test and lower limb muscle strength will be evaluated by using a dynamometer.
  Units: Visual analog scale (VAS 0-10); 0-10 corresponds to the no pain to severe pain.
Neuromuscular Assessment | Baseline, 3 months, 6 months
  For neuromuscular assessment assess the sharp-dull and deep pressure sensation. Units: None
Balance Assessment | Baseline, 3 months, 6 months
  Balance assessment will be measured by Berg balance assessment. Units: Scale 0 to 4, with 4 indicating normal and 0 representing severe impairment
Quality of life Questionnaire | Baseline, 3 months, 6 months, 9 months
  Health related quality of life using a Short-Form 36 general health survey. Units: An arbitrary scale 0 to 100, with higher scores representing better health.
Assessment of PAD Severity | Baseline, 3 months, 6 months, 9 months
  To assess the leg symptoms, participants who are affirmative for the pain in legs or buttock on walking will be characterized by the responses to San Diego Claudication Questionnaire (SDCQ) and Walking Impairment Questionnaire (WIQ)
  Measures: (1) intermittent claudication, (2) leg pain on exertion and rest, (3) atypical exertional leg pain, (4) atypical exertional leg pain/stop, and (5) no exertional pain.
Depressive Symptoms Questionnaire | Baseline, 3 months, 6 months, 9 months
  Depression symptoms will be evaluated using Patient Health Questionnaire-9 (PHQ-9).
  Units: Scores evaluated on a 4-point scale from "not at all" to "nearly every day". PHQ-9 scores of 5, 10, 15, and 20 represented mild, moderate, moderately severe, and severe depression respectively.
24-hour Dietary Recall | Baseline, 3 months, 6 months, 9 months
  Recall of participant's dietary patterns over the past 24 hours from the time of the visit using web-based, Automated Self-Administered 24-hour (ASA24®) Dietary Assessment Tool 2024 Version.
Daily Walking Ability | -7-Baseline, Day 90-97, Day 180-187, Day 270-277
  Steps over a period of 6 days using triaxial pedometer. Units: step counts
Blood Collection and Analysis | Baseline, 3 months, 6 months, 9 months
  White blood cells, red blood cells. Units: Cells per cubic millimeter. Neutrophils, lymphocytes, monocytes, eosinophils, basophils. Units: percent
Blood Collection and Analysis | Baseline, 3 months, 6 months, 9 months
  Sodium, phosphate, chloride, calcium, glucose, creatinine, albumin, ALT and AST Units: mg/dL
Measurement of Carnosine in Blood and Urine | Baseline, 3 months, 6 months, 9 months
  Using mass spectrometry will measure carnosine bioavailability. Units: moles
Measure Angiogenic Cell Population | Baseline, 3 months, 6 months, 9 months
  Flow cytometry: measure angiogenic cell population. Units: Number of cells
Mitochondrial Abundance Measurements | Baseline, 3 months, 6 months, 9 months
  Perform RTPCR to measure expression of different mitochondrial genes. Units: Relative mRNA expression
Measurement of Carnosine in Muscle | Baseline, 6 months
  Using magnetic resonance spectroscopy, will measure carnosine accumulation before and after supplementation.
  Units: millimole.
Measurement of Blood Flow | Baseline, 6 months
  Using magnetic resonance imaging will measure blood flow in the legs. Units: mL/min
Calf Muscle Biopsy | Baseline, 6 months
  Optional muscle biopsy will be obtained by a trained vascular surgeon from the consistent location of medial gastrocnemius of the symptomatic leg using a ¼ inch bore percutaneous biopsy needle.

CONTACTS AND LOCATIONS:
Overall Officials: Shahid Baba, PhD, Principal Investigator — University of Louisville School of Medicine
Locations (3):
- United States (3):
  - University of Louisville School of Medicine, Department of Medicine, Division of Environmental Medicine, Louisville, Kentucky
  - University Surgical Associates, 401 E. Chestnut St, Suite 710, Louisville, Kentucky
  - UofL Physicians - Vascular Surgery Associates, 201 Abraham Flexner Way, Suite 1004, Louisville, Kentucky

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] de Courten B, Jakubova M, de Courten MP, Kukurova IJ, Vallova S, Krumpolec P, Valkovic L, Kurdiova T, Garzon D, Barbaresi S, Teede HJ, Derave W, Krssak M, Aldini G, Ukropec J, Ukropcova B. Effects of carnosine supplementation on glucose metabolism: Pilot clinical trial. Obesity (Silver Spring). 2016 May;24(5):1027-34. doi: 10.1002/oby.21434. Epub 2016 Apr 4. PMID 27040154
- [Background] Vincent KA, Shyu KG, Luo Y, Magner M, Tio RA, Jiang C, Goldberg MA, Akita GY, Gregory RJ, Isner JM. Angiogenesis is induced in a rabbit model of hindlimb ischemia by naked DNA encoding an HIF-1alpha/VP16 hybrid transcription factor. Circulation. 2000 Oct 31;102(18):2255-61. doi: 10.1161/01.cir.102.18.2255. PMID 11056102
- [Background] Hiatt WR, Hoag S, Hamman RF. Effect of diagnostic criteria on the prevalence of peripheral arterial disease. The San Luis Valley Diabetes Study. Circulation. 1995 Mar 1;91(5):1472-9. doi: 10.1161/01.cir.91.5.1472. PMID 7867189
- [Background] Waeckel L, Mallat Z, Potteaux S, Combadiere C, Clergue M, Duriez M, Bao L, Gerard C, Rollins BJ, Tedgui A, Levy BI, Silvestre JS. Impairment in postischemic neovascularization in mice lacking the CXC chemokine receptor 3. Circ Res. 2005 Mar 18;96(5):576-82. doi: 10.1161/01.RES.0000159389.55544.20. Epub 2005 Feb 17. PMID 15718500
- [Background] Gerhardt H, Golding M, Fruttiger M, Ruhrberg C, Lundkvist A, Abramsson A, Jeltsch M, Mitchell C, Alitalo K, Shima D, Betsholtz C. VEGF guides angiogenic sprouting utilizing endothelial tip cell filopodia. J Cell Biol. 2003 Jun 23;161(6):1163-77. doi: 10.1083/jcb.200302047. Epub 2003 Jun 16. PMID 12810700
- [Background] Creager MA, Olin JW, Belch JJ, Moneta GL, Henry TD, Rajagopalan S, Annex BH, Hiatt WR. Effect of hypoxia-inducible factor-1alpha gene therapy on walking performance in patients with intermittent claudication. Circulation. 2011 Oct 18;124(16):1765-73. doi: 10.1161/CIRCULATIONAHA.110.009407. Epub 2011 Sep 26. PMID 21947297
- [Background] Wang GL, Semenza GL. Desferrioxamine induces erythropoietin gene expression and hypoxia-inducible factor 1 DNA-binding activity: implications for models of hypoxia signal transduction. Blood. 1993 Dec 15;82(12):3610-5. PMID 8260699
- [Background] Silvestre JS, Mallat Z, Tedgui A, Levy BI. Post-ischaemic neovascularization and inflammation. Cardiovasc Res. 2008 May 1;78(2):242-9. doi: 10.1093/cvr/cvn027. Epub 2008 Feb 5. PMID 18252762
- [Background] Aicher A, Zeiher AM, Dimmeler S. Mobilizing endothelial progenitor cells. Hypertension. 2005 Mar;45(3):321-5. doi: 10.1161/01.HYP.0000154789.28695.ea. Epub 2005 Jan 17. PMID 15655116
- [Background] Asahara T, Takahashi T, Masuda H, Kalka C, Chen D, Iwaguro H, Inai Y, Silver M, Isner JM. VEGF contributes to postnatal neovascularization by mobilizing bone marrow-derived endothelial progenitor cells. EMBO J. 1999 Jul 15;18(14):3964-72. doi: 10.1093/emboj/18.14.3964. PMID 10406801
- [Background] Forsythe JA, Jiang BH, Iyer NV, Agani F, Leung SW, Koos RD, Semenza GL. Activation of vascular endothelial growth factor gene transcription by hypoxia-inducible factor 1. Mol Cell Biol. 1996 Sep;16(9):4604-13. doi: 10.1128/MCB.16.9.4604. PMID 8756616
- [Background] Ziello JE, Jovin IS, Huang Y. Hypoxia-Inducible Factor (HIF)-1 regulatory pathway and its potential for therapeutic intervention in malignancy and ischemia. Yale J Biol Med. 2007 Jun;80(2):51-60. PMID 18160990
- [Background] Heil M, Schaper W. Influence of mechanical, cellular, and molecular factors on collateral artery growth (arteriogenesis). Circ Res. 2004 Sep 3;95(5):449-58. doi: 10.1161/01.RES.0000141145.78900.44. PMID 15345667
- [Background] Serrano Hernando FJ, Martin Conejero A. [Peripheral artery disease: pathophysiology, diagnosis and treatment]. Rev Esp Cardiol. 2007 Sep;60(9):969-82. doi: 10.1157/13109651. Spanish. PMID 17915154
- [Background] Chez MG, Buchanan CP, Aimonovitch MC, Becker M, Schaefer K, Black C, Komen J. Double-blind, placebo-controlled study of L-carnosine supplementation in children with autistic spectrum disorders. J Child Neurol. 2002 Nov;17(11):833-7. doi: 10.1177/08830738020170111501. PMID 12585724
- [Background] Hobson RM, Saunders B, Ball G, Harris RC, Sale C. Effects of beta-alanine supplementation on exercise performance: a meta-analysis. Amino Acids. 2012 Jul;43(1):25-37. doi: 10.1007/s00726-011-1200-z. Epub 2012 Jan 24. PMID 22270875
- [Background] Parkhouse WS, McKenzie DC, Hochachka PW, Ovalle WK. Buffering capacity of deproteinized human vastus lateralis muscle. J Appl Physiol (1985). 1985 Jan;58(1):14-7. doi: 10.1152/jappl.1985.58.1.14. PMID 3968004
- [Background] Beebe HG, Dawson DL, Cutler BS, Herd JA, Strandness DE Jr, Bortey EB, Forbes WP. A new pharmacological treatment for intermittent claudication: results of a randomized, multicenter trial. Arch Intern Med. 1999 Sep 27;159(17):2041-50. doi: 10.1001/archinte.159.17.2041. PMID 10510990
- [Background] Harwood AE, Smith GE, Cayton T, Broadbent E, Chetter IC. A Systematic Review of the Uptake and Adherence Rates to Supervised Exercise Programs in Patients with Intermittent Claudication. Ann Vasc Surg. 2016 Jul;34:280-9. doi: 10.1016/j.avsg.2016.02.009. Epub 2016 Apr 25. PMID 27126713
- [Background] Treat-Jacobson D, McDermott MM, Bronas UG, Campia U, Collins TC, Criqui MH, Gardner AW, Hiatt WR, Regensteiner JG, Rich K; American Heart Association Council on Peripheral Vascular Disease; Council on Quality of Care and Outcomes Research; and Council on Cardiovascular and Stroke Nursing. Optimal Exercise Programs for Patients With Peripheral Artery Disease: A Scientific Statement From the American Heart Association. Circulation. 2019 Jan 22;139(4):e10-e33. doi: 10.1161/CIR.0000000000000623. No abstract available. PMID 30586765
- [Background] Treat-Jacobson D, McDermott MM, Beckman JA, Burt MA, Creager MA, Ehrman JK, Gardner AW, Mays RJ, Regensteiner JG, Salisbury DL, Schorr EN, Walsh ME; American Heart Association Council on Peripheral Vascular Disease; Council on Cardiovascular and Stroke Nursing; Council on Epidemiology and Prevention; and Council on Lifestyle and Cardiometabolic Health. Implementation of Supervised Exercise Therapy for Patients With Symptomatic Peripheral Artery Disease: A Science Advisory From the American Heart Association. Circulation. 2019 Sep 24;140(13):e700-e710. doi: 10.1161/CIR.0000000000000727. Epub 2019 Aug 26. PMID 31446770
- [Background] McDermott MM, Guralnik JM, Tian L, Zhao L, Polonsky TS, Kibbe MR, Criqui MH, Zhang D, Conte MS, Domanchuk K, Li L, Sufit R, Leeuwenburgh C, Ferrucci L. Comparing 6-minute walk versus treadmill walking distance as outcomes in randomized trials of peripheral artery disease. J Vasc Surg. 2020 Mar;71(3):988-1001. doi: 10.1016/j.jvs.2019.05.058. Epub 2019 Dec 23. PMID 31870756
- [Background] McDermott MM, Dayanidhi S, Kosmac K, Saini S, Slysz J, Leeuwenburgh C, Hartnell L, Sufit R, Ferrucci L. Walking Exercise Therapy Effects on Lower Extremity Skeletal Muscle in Peripheral Artery Disease. Circ Res. 2021 Jun 11;128(12):1851-1867. doi: 10.1161/CIRCRESAHA.121.318242. Epub 2021 Jun 10. PMID 34110902
- [Background] McDermott MM, Spring B, Tian L, Treat-Jacobson D, Ferrucci L, Lloyd-Jones D, Zhao L, Polonsky T, Kibbe MR, Bazzano L, Guralnik JM, Forman DE, Rego A, Zhang D, Domanchuk K, Leeuwenburgh C, Sufit R, Smith B, Manini T, Criqui MH, Rejeski WJ. Effect of Low-Intensity vs High-Intensity Home-Based Walking Exercise on Walk Distance in Patients With Peripheral Artery Disease: The LITE Randomized Clinical Trial. JAMA. 2021 Apr 6;325(13):1266-1276. doi: 10.1001/jama.2021.2536. PMID 33821898
- [Background] Money SR, Herd JA, Isaacsohn JL, Davidson M, Cutler B, Heckman J, Forbes WP. Effect of cilostazol on walking distances in patients with intermittent claudication caused by peripheral vascular disease. J Vasc Surg. 1998 Feb;27(2):267-74; discussion 274-5. doi: 10.1016/s0741-5214(98)70357-x. PMID 9510281
- [Background] Dawson DL, Cutler BS, Meissner MH, Strandness DE Jr. Cilostazol has beneficial effects in treatment of intermittent claudication: results from a multicenter, randomized, prospective, double-blind trial. Circulation. 1998 Aug 18;98(7):678-86. doi: 10.1161/01.cir.98.7.678. PMID 9715861
- [Background] Girolami B, Bernardi E, Prins MH, Ten Cate JW, Hettiarachchi R, Prandoni P, Girolami A, Buller HR. Treatment of intermittent claudication with physical training, smoking cessation, pentoxifylline, or nafronyl: a meta-analysis. Arch Intern Med. 1999 Feb 22;159(4):337-45. doi: 10.1001/archinte.159.4.337. PMID 10030306
- [Background] Peacock JM, Keo HH, Duval S, Baumgartner I, Oldenburg NC, Jaff MR, Henry TD, Yu X, Hirsch AT. The incidence and health economic burden of ischemic amputation in Minnesota, 2005-2008. Prev Chronic Dis. 2011 Nov;8(6):A141. Epub 2011 Oct 17. PMID 22005634
- [Background] Roger VL, Go AS, Lloyd-Jones DM, Adams RJ, Berry JD, Brown TM, Carnethon MR, Dai S, de Simone G, Ford ES, Fox CS, Fullerton HJ, Gillespie C, Greenlund KJ, Hailpern SM, Heit JA, Ho PM, Howard VJ, Kissela BM, Kittner SJ, Lackland DT, Lichtman JH, Lisabeth LD, Makuc DM, Marcus GM, Marelli A, Matchar DB, McDermott MM, Meigs JB, Moy CS, Mozaffarian D, Mussolino ME, Nichol G, Paynter NP, Rosamond WD, Sorlie PD, Stafford RS, Turan TN, Turner MB, Wong ND, Wylie-Rosett J; American Heart Association Statistics Committee and Stroke Statistics Subcommittee. Heart disease and stroke statistics--2011 update: a report from the American Heart Association. Circulation. 2011 Feb 1;123(4):e18-e209. doi: 10.1161/CIR.0b013e3182009701. Epub 2010 Dec 15. PMID 21160056
- [Background] Boakye AA, Zhang D, Guo L, Zheng Y, Hoetker D, Zhao J, Posa DK, Ng CK, Zheng H, Kumar A, Kumar V, Wempe MF, Bhatnagar A, Conklin DJ, Baba SP. Carnosine Supplementation Enhances Post Ischemic Hind Limb Revascularization. Front Physiol. 2019 Jul 2;10:751. doi: 10.3389/fphys.2019.00751. eCollection 2019. PMID 31312142
- [Background] Schon M, Just I, Krumpolec P, Blazicek P, Valkovic L, Aldini G, Tsai CL, De Courten B, Krssak M, Ukropcova B, Ukropec J. Supplementation-induced change in muscle carnosine is paralleled by changes in muscle metabolism, protein glycation and reactive carbonyl species sequestering. Physiol Res. 2023 Mar 8;72(1):87-97. doi: 10.33549/physiolres.934911. Epub 2022 Dec 22. PMID 36545878
- [Background] Caruso J, Charles J, Unruh K, Giebel R, Learmonth L, Potter W. Ergogenic effects of beta-alanine and carnosine: proposed future research to quantify their efficacy. Nutrients. 2012 Jul;4(7):585-601. doi: 10.3390/nu4070585. Epub 2012 Jun 26. PMID 22852051
- [Background] Harris RC, Stellingwerff T. Effect of beta-alanine supplementation on high-intensity exercise performance. Nestle Nutr Inst Workshop Ser. 2013;76:61-71. doi: 10.1159/000350258. Epub 2013 Jul 25. PMID 23899755
- [Background] Hipkiss AR. Energy metabolism, proteotoxic stress and age-related dysfunction - protection by carnosine. Mol Aspects Med. 2011 Aug;32(4-6):267-78. doi: 10.1016/j.mam.2011.10.004. Epub 2011 Oct 15. PMID 22020113
- [Background] Teufel M, Saudek V, Ledig JP, Bernhardt A, Boularand S, Carreau A, Cairns NJ, Carter C, Cowley DJ, Duverger D, Ganzhorn AJ, Guenet C, Heintzelmann B, Laucher V, Sauvage C, Smirnova T. Sequence identification and characterization of human carnosinase and a closely related non-specific dipeptidase. J Biol Chem. 2003 Feb 21;278(8):6521-31. doi: 10.1074/jbc.M209764200. Epub 2002 Dec 6. PMID 12473676
- [Background] Drozak J, Veiga-da-Cunha M, Vertommen D, Stroobant V, Van Schaftingen E. Molecular identification of carnosine synthase as ATP-grasp domain-containing protein 1 (ATPGD1). J Biol Chem. 2010 Mar 26;285(13):9346-9356. doi: 10.1074/jbc.M109.095505. Epub 2010 Jan 22. PMID 20097752
- [Background] Lombardi C, Carubelli V, Lazzarini V, Vizzardi E, Bordonali T, Ciccarese C, Castrini AI, Dei Cas A, Nodari S, Metra M. Effects of oral administration of orodispersible levo-carnosine on quality of life and exercise performance in patients with chronic heart failure. Nutrition. 2015 Jan;31(1):72-8. doi: 10.1016/j.nut.2014.04.021. Epub 2014 May 10. PMID 25287762
- [Background] Criqui MH, Aboyans V. Epidemiology of peripheral artery disease. Circ Res. 2015 Apr 24;116(9):1509-26. doi: 10.1161/CIRCRESAHA.116.303849. PMID 25908725
- [Background] Annex BH. Therapeutic angiogenesis for critical limb ischaemia. Nat Rev Cardiol. 2013 Jul;10(7):387-96. doi: 10.1038/nrcardio.2013.70. Epub 2013 May 14. PMID 23670612